CLINICAL TRIAL: NCT03846245
Title: AlfaAge: Cross-sectional Study for the Identification of Blood Biomarkers in Healthy Young and Old Individuals
Brief Title: Cross-sectional Study for the Identification of Blood Biomarkers in Healthy Young and Old Individuals
Acronym: AlfaAge
Status: Completed | Type: Observational
Sponsor: Barcelonabeta Brain Research Center, Pasqual Maragall Foundation (Other)
Collaborators: Göteborg University (Other)
Responsible Party: Sponsor
Other Study IDs: AlfaAge/BBRC2018
Record Dates: First submitted 2019-02-18; First posted 2019-02-19 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Aging

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma and serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Young adults group: Cognitively unimpaired 18-25 years old
  Interventions: Other: No intervention
- Old adults group: Cognitively unimpaired >= 70 years old
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Ageing is clearly the most important risk factor for AD and other dementias but, despite the amount of evidence supporting this fact, the exact mechanism that link ageing and AD is still unknown and, up to now, potential therapies for AD by targeting ageing have been poorly explored. This study aims to provide a better understanding of the link between ageing and AD by means of measuring in human blood those factors that have been found to be 'pro-youthful' (GDF-11, CSF2, TIMP-2, oxytocin) or 'pro-aging' (CCL2, CCL11, CCL19, Haptoglobine, B2-microglobuline) in experimental animal models, but have not been comprehensively studied in humans.

In this proof-of-concept study these blood factors in extreme groups of age, namely young adults (18-25 yo) and old adults (≥70 yo) will be measured and the hypothesis of whether the 'pro-youthful' and 'pro-ageing' blood factors change throughout age tested. In order to include a wider range of age, human umbilical cord blood and plasma from teenagers (which is already available from a previous study) will also be included.

The ultimate goal of this study is to select the more promising blood factors and obtain data on the effect size of the differences that may allow us in the future to design a larger study.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between 18 and 25 years (young adults group) or older than 70 for persons at the time of inclusion (old adults group).
2. Subjects with no subjective cognitive complaints.
3. Individuals interested in participating in the study who fully understand all the procedures that will be performed.
4. Explicit participant agreement to undergo all the study procedures, which encompass:

   1. Collection of basic demographic data.
   2. Collection of a blood sample.
5. Give informed consent and agree that no data resulting from the study (which is no clinically relevant) will be given to the participant

Exclusion Criteria:

1. No signs of subjective cognitive impairment.
2. Any significant systemic illness or unstable medical condition which could lead to difficulty complying with the protocol. Including: auditive and visual impairment, renal insufficiency under hemodialysis treatment, hepatic cirrhosis, chronic pneumopathy under oxygen therapy, solid organ transplantation, fibromyalgia, active oncologic disease under treatment (excluding localized tumours).
3. Any significant major psychiatric illness (following DSM-IV diagnosis manual) o diseases that interfere with cognitive function (including major depression disorder, bipolar disorder, schizophrenia).
4. Acquired brain injury: brain traumatic injury with parenchymal or extra-axial macroscopic injury, large vessel ischemic stroke or hemorrhagic stroke, brain tumors or other conditions that may cause acquired brain injury (brain radio- or chemotherapy).
5. Parkinson's disease, epilepsy under treatment and with frequent seizures (>1 /month) in the last year, multiple sclerosis or any other neurodegenerative disease.
6. Researcher criteria: individuals that have any condition which, under researcher's view, could lead to difficulty complying with the protocol.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Cognitively unimpaired subjects
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2019-05-03 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Concentration of CCL2 | at inclusion
  Differences in the concentration of CCL2 between age groups
Concentration of CCL11 | at inclusion
  Differences in the concentration of CCL11 between age groups
Concentration of CCL19 | at inclusion
  Differences in the concentration of CCL19 between age groups
Concentration of Haptoglobin | at inclusion
  Differences in the concentration of Haptoglobin between age groups
Concentration of B2-microglobulin | at inclusion
  Differences in the concentration of B2-microglobulin between age groups
Concentration of TIMP2 | at inclusion
  Differences in the concentration of TIMP2 between age groups
Concentration of CSF2 | at inclusion
  Differences in the concentration of CSF22 between age groups
Concentration of GDF11 | at inclusion
  Differences in the concentration of GDF11 between age groups
Concentration of oxytoxin | at inclusion
  Differences in the concentration of oxytoxin between age groups

CONTACTS AND LOCATIONS:
Locations (1):
- Barcelonabeta Brain Research Center, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No